CLINICAL TRIAL: NCT06149416
Title: Post-Launch Hypoxia Clinical Study Protocol for Reprocessed Masimo RD SET Pulse Oximeters With Motion
Brief Title: SpO2 Accuracy of Noninvasive Pulse Oximeter Sensor With Motion Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Sustainability Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRD10351
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental Arms (Experimental): Experimental: Healthy adult participants All participants are enrolled in the test group and receive the noninvasive adhesive reprocessed pulse oximeter sensors
  Interventions: Device: Experimental Masimo RD SET SpO2 Adhesive Sensors

INTERVENTIONS:
Device: Experimental Masimo RD SET SpO2 Adhesive Sensors — Masimo RD SET SpO2 Adhesive Sensors, Adult (4000 Adt), Adult & Neonate (4003 Neo)

SUMMARY:
The purpose of this clinical study is to validate the SpO2 accuracy of the Stryker Sustainability Solutions pulse oximetry sensors during motion conditions over the range of 70 -100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry during conditions in which the subject is moving. The end goal is to provide supporting documentation for the SpO2 accuracy validation of the reprocessed sensors with motion indications.

DETAILED DESCRIPTION:
In this study, the level of oxygen within the blood will be reduced in a controlled manner by reducing the concentration of oxygen the study volunteer breathes. The accuracy of a noninvasive pulse oximeter sensor will be assessed by comparison to the oxygen saturation measurements from a laboratory blood gas analyzer.

A machine will be used to induce motions of 20 mm during testing at a sine rate of 2Hz, 3Hz, and 4Hz. A third motion moves the arm a random distance of 0 to 30mm at a random speed up to 5Hz.

It is required that the Accuracy Root Mean Square (ARMS) performance of the Stryker pulse oximetry sensors will meet a specification of +/-3% with a target of +/-3% or better in motion conditions for the range of 70 - 100% SaO2 (typically, saturation is determined once with air breathing and then at three or six levels, e.g. 94%, 90%, 85%, 80%, 75% and 70% or 95%, 85% and 75% saturation for about 30-60 seconds or 60-90 seconds at each level), thereby demonstrating an acceptable SpO2 accuracy performance specification. This study should utilize a three level structure (95%, 85% and 75%).

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female, aged ≥18 and <50
* The subject is in good general health with no evidence of any medical problems.
* The subject is fluent in both written and spoken English
* The subject has provided informed consent and is willing to comply with the study procedures

Exclusion Criteria:

The subject is obese (BMI>30)

* The subject has a known history of heart disease, lung disease, kidney or liver disease
* Diagnosis of asthma, sleep apnea, or use of CPAP
* Subject has diabetes
* Subject has a clotting disorder
* The subject a hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation
* The subject has any other serious systemic illness
* The subject is a current smoker
* Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators would interfere with the sensors working correctly
* The subject has a history of fainting or vasovagal response
* The subject has a history of sensitivity to local anesthesia
* The subject has a diagnosis of Raynaud's disease
* The subject has unacceptable collateral circulation based on exam by the investigator (Allen's test)
* The subject is pregnant, lactating or trying to get pregnant
* The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures
* The subject has any other condition, which in the opinion of the investigators would make them unsuitable for the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2023-05-27 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2023-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bickler, MD, PhD, Principal Investigator — UCSF Hypoxia Research Laboratory
Locations (1):
- UCSF Hypoxia Research Laboratory, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Adult Participants: Experimental: Healthy adult participants All participants are enrolled in the test group and receive the noninvasive adhesive reprocessed pulse oximeter sensors
  Experimental Masimo RD SET SpO2 Adhesive Sensors: Masimo RD SET SpO2 Adhesive Sensors, Adult (4000 Adt), Adult & Neonate (4003 Neo)
Period: Overall Study
Arm/Group | Healthy Adult Participants
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Adult Participants
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5
  Black | 2
  Asian | 2
  Hispanic | 0
  Multiethnic | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor by Comparing SpO2 Percent Blood Oxygen Saturation to SaO2 Percent Blood Oxygen Saturation Utilizing Arms Calculation Calculation [Time Frame: 1 - 5 Hours]
Description: The outcome of this study is the accuracy of the SpO2 (percent oxygen saturation by pulse oximetry) measured by the Reprocessed Oximeter pulse oximetry sensors during motion conditions over the range of 70 - 100% saturation compared to SaO2 (percent oxygen saturation by co-oximetry from blood samples) from arterial blood samples. The accuracy is calculated using the Arms error between measured SpO2 and reference SaO2. The Arms must meet the 3% specification for each reprocessed pulse oximetry sensor style. Standard deviation of the differences is computed as the precision. Square root of the sum of the squares of bias and precision is computed as the Arms Error value.
Time Frame: 1 - 5 hours
Measure: Number; unit: Root Mean Square Error (%)
Groups:
- Masimo RD SET SpO2 Adhesive Sensors: Adult (4000 Adt), Adult & Neonate (4003): Experimental: Healthy adult participants All participants are enrolled in the test group and receive the noninvasive adhesive reprocessed pulse oximeter sensors
Arm/Group | Masimo RD SET SpO2 Adhesive Sensors: Adult (4000 Adt), Adult & Neonate (4003)
Number analyzed (Participants) | 11
Root Mean Square Error (%)
  Device 1 4000-Adt Accuracy | 1.84
  Device 2 4003-Neo Accuracy | 2.33

ADVERSE EVENTS:
Time Frame: 2 Days
Arm/Group | Healthy Adult Participants
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT06149416/Prot_SAP_ICF_000.pdf